CLINICAL TRIAL: NCT01481922
Title: Should Physicians Use a 24 Gauge Spinal Needle Instead of a 22 Gauge When Performing a Lumbar Puncture ? A Randomized Controlled Trial.
Brief Title: What Needle Diameter Should Physician Use When They Perform Lumbar Puncture ? A Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: funding: McGill Emergency Medicine 2010 Grant Competition (Unknown)
Responsible Party: Principal Investigator, Liam Durcan, MD, FRCPc, Neurologist-in-Chief, Montreal Neurological Hospital Interim Clinical Director, Neurology, McGill University Health Center, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NEU-11-001
Record Dates: First submitted 2011-11-15; First posted 2011-11-30 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Post-lumbar Puncture Headache; Backache
Keywords: Lumbar puncture; Flow rate; Backache; Pain; Undifferentiated headache; Post-lumbar puncture headache
MeSH Terms: conditions — Post-Dural Puncture Headache; Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whitacre 22 gauge (Active Comparator): lumbar puncture performed with a Whitacre 22 gauge (BD)
  Interventions: Device: whitacre 22 gauge
- Whitacre 24 gauge (Experimental): lumbar puncture performed with a Whitacre 24 gauge (BD)
  Interventions: Device: whitacre 24 gauge

INTERVENTIONS:
Device: whitacre 24 gauge — Whitacre 24 gauge spinal needle 3 inches 1/2. Manufactured by Becton Dickinson
  Other Names: Product number: 405133
  Arms: Whitacre 24 gauge
Device: whitacre 22 gauge — Whitacre 22 gauge spinal needle 3 inches 1/2 manufactured by Becton Dickinson
  Other Names: product number 405010
  Arms: Whitacre 22 gauge

SUMMARY:
This study is intended to help guide the choice of needle diameter when performing a lumbar puncture.

Smaller spinal needles have been shown to decrease rate of adverse events such as post-lumbar puncture headache and hearing loss.

The main drawback to using smaller needles is diminished flow rate; some textbooks recommend using needles no smaller than 22 gauge because of the slow flow rate though others recommend smaller needles, namely 22-24 gauge.

Some authors have described a successful use of spinal needles as small as 25 gauge when performing a lumbar puncture.

The investigators do not believe that the flow-rate difference between 22 and 24 gauge needles is significant enough to justify using the larger needles.

The investigators trial will compare the Whitacre 22 gauge and Whitacre 24 gauge needles for flow rate, and incidence of the known complications of pain during procedure and backache at 8 and 15 days post-procedure.

The investigators will also look at whether smaller needles are associated with less pain during the procedure and less backache the next 2 weeks after the procedure.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blinded clinical trial is to assess whether a 24 gauge spinal needle can provide an acceptable flow rate of cerebrospinal fluid (CSF) when compared to the traditionally used 22 gauge needle.

Smaller needles, according to The Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology are 'associated with reduced frequency of post-lumbar puncture headache (Level A recommendation).'

Given that flow rate of CSF is the limiting factor when choosing a spinal needle gauge, two previous studies have compared various needle sizes for adequacy of flow. These studies, however, have important limitations and have not led to a clear consensus in clinical practice. For instance, one study used a 0,9 % solution of sodium chloride at room temperature, the other used an 'artificial CSF solution' of unknown viscosity and nature.

Patients referred to the neurological day center of the Montreal Neurological Institute/Hospital for lumbar puncture will be recruited to the study. Participants will be randomized to have the puncture with a Whitacre 22 or 24 gauge needle.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (>= 18 years old) referred at the Neurological Day Center to get a lumbar puncture

Exclusion Criteria:

* Contraindication to get a lumbar puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Time to collect 5 ml of CSF | after 5 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 5 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 5ml, the time will be adjusted accordingly to reflect collection of exactly 5ml.

SECONDARY OUTCOMES:
Time to collect 7 ml of CSF | after 7 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 7 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 7 ml, the time will be adjusted accordingly to reflect collection of exactly 7 ml.
Time to collect 8 ml of CSF | after 8 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 8 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 8 ml, the time will be adjusted accordingly to reflect collection of exactly 8 ml.
Time to collect 9 ml of CSF | after 9 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 9 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 9 ml, the time will be adjusted accordingly to reflect collection of exactly 9 ml.
Time to collect 10 ml of CSF | after 10 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 10 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 10 ml, the time will be adjusted accordingly to reflect collection of exactly 10 ml.
Time to collect 6 ml of CSF | after 6 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 6 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 6 ml, the time will be adjusted accordingly to reflect collection of exactly 6 ml.
Time to collect 11 ml of CSF | after 11 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 11 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 11 ml, the time will be adjusted accordingly to reflect collection of exactly 11 ml.
Time to collect 12 ml of CSF | after 12 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 12 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 12 ml, the time will be adjusted accordingly to reflect collection of exactly 12 ml.
Time to collect 13 ml of CSF | after 13 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 13 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 13 ml, the time will be adjusted accordingly to reflect collection of exactly 13 ml.
Time to collect 15 ml of CSF | after 15 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 15 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 15 ml, the time will be adjusted accordingly to reflect collection of exactly 15 ml.
Backache first 8 days after the lumbar puncture (LP) | Assessed at 8 days after the LP
  The presence of backache since the LP will be assessed by phone call by a blinded research assistant.
Severity of backache first 8 days after the LP | Assessed at 8 days after the LP
  The severity of the backache (when present) will be assessed at 8 days by a phone call by a blinded research assistant.
  A numerical rating scale will be used (0-10)
Severity of backache first 15 days after the LP | Assessed at 15 days after the LP
  The severity of the backache (when present) will be assessed at 15 days by a phone call by a blinded research assistant.
  A numerical rating scale will be used (0-10)
Backache first 15 days after the LP | Assessed at 15 days after the LP
  The presence of backache since the LP will be assessed by phone call by a blinded research assistant.
Post-lumbar puncture headache (PLPH) at 8 days | 8 days after the LP
  The presence of PLPH since the LP will be assessed by phone call by a blinded research assistant. The International Headache Society definition of PLPH will be used.
Post-lumbar puncture headache (PLPH) at 15 days | 15 days after the LP
  The presence of PLPH since the LP will be assessed by phone call by a blinded research assistant. The International Headache Society definition of PLPH will be used.
Severity of the post-lumbar puncture headache (PLPH) at 8 days | 8 days after the LP
  The severity of PLPH (when present) will be assessed by phone call by a blinded research assistant. A numerical rating scale (0-10) will be used.
Severity of the post-lumbar puncture headache (PLPH) at 15 days | 15 days after the LP
  The severity of PLPH (when present) will be assessed by phone call by a blinded research assistant. A numerical rating scale (0-10) will be used.
Time to get CSF | During the LP
  The time required to get a successful LP will be measured. Start time (T=0s) will be the first contact of the spinal needle with the skin. Stop time will be when the first drop of CSF drips out of the needle hub
Extra time patients are willing to spend - part 1 | immediately after the LP
  Patients will be asked right after the LP by a blinded research assistant how much more time they would have been willing to spend for an LP if it could reduce the rate of PLPH and hearing loss
Extra time patients are willing to spend - part 2 | 8 days after LP
  Patients will be asked 8 days after the LP by a blinded research assistant how much more time they would have been willing to spend for an LP if it could reduce the rate of PLPH and hearing loss Subgroup analysis will be done for patient who developed PLPH
Extra time patients willing to spend - part 3 | 15 days after LP
  Patients will be asked 15 days after the LP by a blinded research assistant how much more time they would have been willing to spend for an LP if it could reduce the rate of PLPH and hearing loss Subgroup analysis will be done for patient who developed PLPH
Pain related to LP | Immediately after LP
  The severity of the pain related to the LP will be assessed by a blinded research assistant using a visual analogue scale (0-10)
Number of attempts | during the LP
  The number of attempts before collection of CSF is successful will be recorded
Medical attention for PLPH | at 15 days
  The need for patients to get medical assistance regarding a PLPH will be recorded (as defined by: a visit to health-care provider, admission to hospital, or a phone call to a health-care provider). This will be determined by a phone call at 15 days by a blinded research assistant.
Medical attention for backache | at 8 days
  The need for patients to get medical assistance regarding a backache will be recorded (as defined by: a visit to health-care provider, admission to hospital, or a phone call to a health-care provider). This will be determined by a phone call at 8 days by a blinded research assistant.
Medical attention for backache | at 15 days
  The need for patients to get medical assistance regarding a backache will be recorded (as defined by: a visit to a health-care provider, admission to hospital, or a phone call to a health-care provider). This will be determined by a phone call at 15 days by a blinded research assistant.
Medical treatment for PLPH | 8 days
  Patient will be asked by phone by a blinded research assistant if they received a medical treatment for their PLPH (eg. analgesics).
Medical treatment for PLPH | 15 days
  Patient will be asked by phone by a blinded research assistant if they received a medical treatment for their PLPH (eg. analgesics)
Medical treatment for backache | 8 days
  Patient will be asked by phone by a blinded research assistant if they received a medical treatment for their backache(eg. analgesics)
Medical treatment for backache | 15 days
  Patient will be asked by phone by a blinded research assistant if they received a medical treatment for their backache(eg. analgesics)
Epidural blood patch for PLPH | at 8 days
  Patients will be asked by phone by a blinded research assistant if they received an epidural blood patch for PLPH.
Epidural blood patch for PLPH | at 15 days
  Patients will be asked by phone by a blinded research assistant if they received an epidural blood patch for PLPH.
Undifferentiated headache at 8 days | 8 days after the LP
  The presence of any headache since the LP will be assessed by phone call by a blinded research assistant.
Undifferentiated headache at 15 days | 15 days after the LP
  The presence of any headache since the LP will be assessed by phone call by a blinded research assistant.
Hearing loss | 8 days after LP
  The presence of subjective hearing loss will be recorded at 8 days by a phone call by a blinded research assistant
Hearing loss | 15 days after LP
  The presence of subjective hearing loss will be recorded at 8 days by a phone call by a blinded research assistant
Time to collect 14 ml of CSF | after 14 ml of CSF is retrieved
  Time 0 will be when the first drop of CSF emerges from the needle hub. Time stops when 14 ml of CSF is retrieved (last drop dripping out of the needle hub) Volume will be confirmed by a blinded research assistant. In the event that the volume differs slightly from 14 ml, the time will be adjusted accordingly to reflect collection of exactly 14 ml.
Medical attention for PLPH | at 8 days
  The need for patients to get medical assistance regarding a PLPH will be recorded (as defined by: a visit to health-care provider, admission to hospital, or a phone call to a health-care provider). This will be determined by a phone call at 8 days by a blinded research assistant.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Durcan, MD, FRCP(c), Principal Investigator — Montreal Neurological Hospital and Institute, McGill University
Locations (1):
- Montreal Neurological Hospital and Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Armon C, Evans RW; Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Addendum to assessment: Prevention of post-lumbar puncture headaches [RETIRED]: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2005 Aug 23;65(4):510-2. doi: 10.1212/01.wnl.0000173034.96211.1b. PMID 16116106
- [Background] Abouleish E, Mitchell M, Taylor G, Miller H, Warters D, Rashad MN. Comparative flow rates of saline in commonly used spinal needles including pencil-tip needles. Reg Anesth. 1994 Jan-Feb;19(1):34-42. PMID 8148292
- [Background] Carson D, Serpell M. Choosing the best needle for diagnostic lumbar puncture. Neurology. 1996 Jul;47(1):33-7. doi: 10.1212/wnl.47.1.33. PMID 8710120